CLINICAL TRIAL: NCT02903810
Title: A Phase I/II Study of Combination Transfer of αCD19-TCRz-41BB and αCD22-TCRz-41BB Chimeric Antigen Receptor T-Cells in Patients With Refractory or Recurrent CD19/22+ B-lineage Leukemia/Lymphoma
Brief Title: Combination Transfer of αCD19-TCRz-41BB and αCD22-TCRz-41BB CAR-T Cells for B-cell Hematologic Malignancy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Jiang Cao, Director of Hematology, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XZCJ20160001
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Hematopoietic/Lymphoid Cancer
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mixed CAR-T Transfer (Experimental): All subjects will be infused with αCD19-TCRz-41BB and αCD22-TCRz-41BB CAR-T cells in equal number
  Interventions: Biological: Mixed CAR-T Transfer

INTERVENTIONS:
Biological: Mixed CAR-T Transfer — All subjects will be infused with αCD19-TCRz-41BB and αCD22-TCRz-41BB CAR-T cells in equal number

SUMMARY:
Clinical study of CD19 CAR-T in the treatment of blood and lymphatic system tumor has been achieved a breakthrough. The main solution in clinical research is to use CD19 CAR-T infusion alone. Because of the heterogeneity of the tumor, the patient often carries tumor cells with CD19 deficient but other positive target antigens (such as CD22). Specifically removal of CD19 positive tumor cells in CAR-T treatment, CD19 negative tumor cells or tumor cells which carry other target antigens would amplify with extra free space released at the same time, resulting in the relapse of tumors of heterogeneities. In order to effectively control the recurrence, CAR-T treatment scheme specific for several target antigens was presented and verified. However treatment with the sequential infusion of different target specific CAR-T cells, the window period between two times infusions may be the opportunity for the tumor recurrence of heterogeneity; and bispecific CAR-T has also been reported only one CAR can be fully functioned. In order to avoid these problems, this topic puts forward for the first time in the international with a treatment scheme of an equal amount of infusion of CD19-41BB and CD22-41BB two Car-T in the treatment of refractory hematologic malignancies. We expect the treatment is more effective in eliminating tumor burden, and also can inhibit the recurrence of tumor heterogeneity at the same time.

DETAILED DESCRIPTION:
To determine:

Primary Outcome Measure:

* Safety (incidence of adverse events defined as dose-limited toxicity)

Secondary Outcome Measures:

* Survival of CAR T cells in circulation measured by flow cytometry and qPCR
* Overall complete remission rate
* Tissue infiltration of transferred CAR-T cells
* In vitro killing potential of infiltrated CAR-T cells
* Phenotype of infused CAR-T cells

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 70 Years, Male and female
* Expected survival > 12 weeks
* Performance score 0-2
* Histologically confirmed as CD19/22-positive lymphoma/leukemia and who meet one of the following conditions; Patient receive at least 2-4 prior combination chemotherapy regimens (not including single agent monoclonal antibody therapy) and fail to achieve CR; or have disease recurrence; or not eligible for allogeneic stem cell transplantation; or disease responding or stable after most recent therapy but refused further treatment; Disease recurrence after stem cell transplantation; Diagnosis as lymphoma, but refuse conventional treatment such as chemotherapy, radiation, stem cell transplantation and monoclonal antibody therapy
* Creatinine < 2.5 mg/dl;
* ALT/AST < 3x normal;
* Bilirubin < 2.0 mg/dl;
* Adequate venous access for apheresis, and no other contraindications for leukapheresis;
* Take contraceptive measures before recruit to this trial;
* Written voluntary informed consent is given.

Exclusion Criteria:

* Patients with symptoms of central nervous system
* Accompanied by other malignant tumor
* Active hepatitis B or C, HIV infection
* Any other diseases could affect the outcome of this trial
* Suffering severe cardiovascular or respiratory disease
* Poorly controlled hypertension
* A history of mental illness and poorly controlled
* Taking immunosuppressive agents within 1 week due to organ transplantation or other disease which need long-lasting administration
* Occurrence of unstable pulmonary embolism, deep vein thrombosis, or other major arterial/venous thromboembolic events 30 days prior to assignment
* Reaching a steady dose if receiving anticoagulant therapy before assignment
* Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
* Pregnant or lactating women
* Subject suffering disease affects the understanding of informed consent or comply with study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Safety (incidence of adverse events defined as dose-limited toxicity) | 30 days

SECONDARY OUTCOMES:
Survival of CAR T cells in circulation measured by flow cytometry and qPCR | 1 years
Overall complete remission rate | 8 weeks
Tissue infiltration of transferred CAR-T cells | 1 years
In vitro killing potential of infiltrated CAR-T cells | 1 years
Phenotype of infused CAR-T cells | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Cao, Doctor, Principal Investigator — Xuzhou Medical University
Locations (1):
- XuZhou Medical University, Xuzhou, Jiangsu, China